CLINICAL TRIAL: NCT04361045
Title: Randomized Control Trial of Online Mental Health Promotion Program for University Students
Brief Title: StriveWeekly: Self-Guided Online Intervention for Anxiety, Depression, and Stress in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Leslie Rith-Najarian, PhD, Postdoctoral Fellow and Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-000761
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Depressive Symptoms; Stress, Psychological
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): Participants in this condition were delivered 8 weeks of online intervention modules and then were invited to complete a posttest survey.
  Interventions: Behavioral: StriveWeekly
- Waitlist Condition (No Intervention): Participants in this condition received no intervention content nor communications for 8 weeks and then were invited to complete a posttest survey.

INTERVENTIONS:
Behavioral: StriveWeekly — The intervention (app.striveweekly.com) delivered eight modules: introduction module, six skills modules, and wrap-up module. The two program "brand name" versions had identical content, but different aesthetic schemes. Modules were released week-by-week, and participants self-guided through content. To facilitate skills practice, every module was accompanied by: a weekly intro email and reminder emails; an "extras" section for tips/suggestions; and a weekly prize drawing. The "Dashboard" section of the intervention displayed user progress. The "Campus" section of this dashboard provided: campus-specific announcements; referrals to relevant campus wellness resources; and an anonymous livestream of all campus users' activity.
  Strategies/skills included: Psychoeducation; Self-monitoring; Behavioral activation; Cognitive restructuring; Sleep hygiene; Time management; Interpersonal avoidance exposures; Physical exercise; Mindfulness; Maintenance planning.
  Other Names: The Happiness Challenge; ReBoot Camp
  Arms: Intervention Condition

SUMMARY:
This study was a randomized controlled trial of an original online mental health promotion program. This study aimed to: 1) establish program effectiveness by examining symptom change between conditions and 2) examine predictors of symptom change. The program was previously tested in open trial feasibility study by the same Principal Investigator and has since been rebuilt as informed by feasibility findings and participant qualitative feedback.

Participants were randomly assigned to either a waitlist condition or eight weeks of the intervention condition. Baseline, posttest, and follow-up electronic surveys collected self-reported symptoms of stress, anxiety, and depression. Motivational variables were also assessed at baseline and then tested as moderators of intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* enrolled as a student at UCLA (Fall 2017 - Winter 2018)

Exclusion Criteria:

* concurrent enrollment in a similar online anxiety and depression treatment study on campus
* invalid data reporting (e.g., straight-lined responses to surveys) -- post hoc exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1631 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS-21) | [Time Frame: Baseline to Posttest (~8 weeks)]
  This 21-item self-report measure assesses symptoms of depression, anxiety, and stress. Individual items are rated 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time), with total scores ranging 0 - 63. Lower scores at posttest relative to baseline indicate improvement.

SECONDARY OUTCOMES:
Program Adherence | [Time Frame: Baseline to Posttest (~8 weeks)]
  This outcome was assessed based on number of modules with 1+ skills practice log. Skills practice logs were recorded as behavioral data, stored within the online platform's database of user account activity.
Program Satisfaction | Posttest (~8 weeks)
  This 5-item measure was adapted from the Client Satisfaction Questionnaire. Individual items are rated 1 (Poor) to 4 (Excellent), with total scores ranging 5 - 20. Higher scores indicate more satisfaction.

OTHER OUTCOMES:
Subjective Happiness Scale | [Time Frame: Baseline to Posttest (~8 weeks)]
  This 4-item self-report measure assesses subjective happiness. Individual items are rated 1 to 7, with total scores ranging 4 - 28. Higher scores at posttest relative to baseline indicate improvement.
Patient Health Questionnaire-9 | [Time Frame: Baseline to Posttest (~8 weeks)]
  This 9-item self-report measure assesses symptoms of major depressive disorder. Individual items are rated 0 (Not at all) to 3 (Nearly every day), with total scores ranging 0 - 27. Lower scores at posttest relative to baseline indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Chavira, PhD, Study Chair — University of California, Los Angeles; Leslie Leslie, PhD, Principal Investigator — Harvard University
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Hanano M, Rith-Najarian L, Gong-Guy E, Chavira D. Motivational Variables as Moderating Effects of a Web-Based Mental Health Program for University Students: Secondary Analysis of a Randomized Controlled Trial. JMIR Form Res. 2024 Jul 3;8:e56118. doi: 10.2196/56118. PMID 38959024
- [Derived] Rith-Najarian LR, Gong-Guy E, Flournoy JC, Chavira DA. Randomized controlled trial of a web-based program for preventing anxiety and depression in university students. J Consult Clin Psychol. 2024 Jan;92(1):1-15. doi: 10.1037/ccp0000843. Epub 2023 Sep 28. PMID 37768633
- [Derived] Hanano M, Rith-Najarian L, Boyd M, Chavira D. Measuring Adherence Within a Self-Guided Online Intervention for Depression and Anxiety: Secondary Analyses of a Randomized Controlled Trial. JMIR Ment Health. 2022 Mar 28;9(3):e30754. doi: 10.2196/30754. PMID 35343901

DOCUMENTS (1):
  • Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT04361045/ICF_000.pdf